CLINICAL TRIAL: NCT03092635
Title: Pilot Study of Pharmacologic Manipulation of AGE (Advanced Glycation Endproducts) Levels in ER+, Metastatic Breast Cancer Patients Receiving Endocrine Therapy
Brief Title: AGE Levels in ER+ Metastatic Breast Cancer Patients Receiving Endocrine Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Original principal investigator departed institution and concluded the study upon departure.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102560
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OPC (Experimental): During weeks 1- 12, subjects will take one OPC tablet in the morning and in the evening, about 12 hours apart.
  Interventions: Drug: OPC

INTERVENTIONS:
Drug: OPC — OPC is a derivative of grape seed extract

SUMMARY:
The purpose of this study is to look at the effects that the study drug (OPC) has on AGE levels in patients with ER+ metastatic breast cancer.

DETAILED DESCRIPTION:
AGEs are a type of metabolite, or substance, found in the food. The AGE content in food is determined by the types of food you eat and also how you prepare your food. The researchers helping conduct this study have found a potential link between AGE levels and cancer. The purpose of this study is to see if certain drug (OPC) has an effect on the AGE levels in your blood and to see if those AGE levels have an effect on your cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must have ER+ breast cancer
* Metastatic disease; protocol does allow for bone-only disease
* Must be receiving endocrine therapy
* Must have completed at last 2 months of current endocrine therapy prior to registration
* Must have adequate hematologic, renal and hepatic function
* Prior/concurrent radiation therapy is allowed
* Prior chemotherapy is allowed, but last dose must have been at least 2 months prior to enrollment
* May have diabetes, but must not be taking metformin
* Must be able to swallow and retain oral medication
* Performance status of 0-2
* Treated stable brain metastases are allowed, as long as patient does not require steroids or anti-seizure medications
* Must be informed of the investigational nature of this study and must have the ability to sign informed consent.

Exclusion Criteria:

* Known allergy to grapes or grape seed
* More than two prior endocrine therapy regimens for the treatment of metastatic ER+ breast cancer.
* Concurrent use of restricted agents outlined in section 4.5.
* History of alcohol abuse within 2 years of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
AGE level reduction | 85 days
  The primary objective is to determine if the test agents are able to reduce AGE levels by at least 30% in th 50% or more of test subjects.

SECONDARY OUTCOMES:
Correlation between AGE level and changes to BMI | 85 days
  Changes in AGE levels and BMI will be described using graphs and other models.
Correlation between AGE level and insulin resistance (HOMA-IR) | 85 days
  Changes in AGE levels and HOMA-IR will be described using graphs and other models.
Correlation between AGE level and A1C | 85 days
  Changes in AGE levels and A1C will be described using graphs and other models.
Correlation between AGE level and lipids | 85 days
  Changes in AGE levels and lipids will be described using graphs and other models.
Correlation between AGE level and diet | 85 days
  Changes in AGE levels and diet will be described using graphs and other models. Diet will be assessed by using the NIH "Eating at America's Table Study Quick Food Scan" and the NCI "Quick Food Scan"
Correlation between AGE level and quality of life | 85 days
  Measured by FACT-B quality of life questionnaire
Correlation between AGE level and plasma IL6 | 85 days
  Changes in AGE levels and IL6 will be described using graphs and other models.
Correlation between AGE level and leptin | 85 days
  Changes in AGE levels and leptin will be described using graphs and other models.
Correlation between AGE level and c-reactive protein (CRP) | 85 days
  Changes in AGE levels and CRP will be described using graphs and other models.
Correlation between AGE level and malondialdehyde (MDA) | 85 days
  Changes in AGE levels and MDA will be described using graphs and other models.
Correlation between AGE level and oxLDLs (low density lipoprotein) | 85 days
  Changes in AGE levels and oxLDLs will be described using graphs and other models.
Correlation between AGE level and sRAGE (soluble receptor for AGE) | 85 days
  Changes in AGE levels and sRAGE will be described using graphs and other models.
Frequency of adverse events as assessed by CTCAE v. 4 | 85 days
  Toxicities will be tabulated by type, grade and the visit at which they occurred.
Tumor response to treatment as assessed by RECIST 1.1 or MD Anderson criteria | 85 days
  The anti-tumor response will be measured by comparing baseline and post-treatment imaging using RECIST 1.1 or MD Anderson criteria for bone only disease.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lilly, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No